CLINICAL TRIAL: NCT00911092
Title: Study of Predictive Proteomic Factors of the Response to Exclusive Concomitant Radiochemotherapy in Oesophageal Cancer
Brief Title: Predictive Proteomic Factors of the Response to Concomitant Radiochemotherapy in Esophageal Cancer
Acronym: COL06-13
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2006-13; NCT00932815 (obsolete NCT alias)
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Esophageal Cancer
Keywords: Oesophageal cancer; exclusive concomitant radiochemotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Blood Specimen Collection; Radiation; Drug Therapy; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sampling — Before any study treatment, 14 days after radiotherapy, 15 weeks after radiotherapy
Radiation: Radiation — Week 1 to week 5-6 1.8-2 Gys/fraction, 5 days a week for a total of 5 to 6 weeks
Drug: Chemotherapy (Fluorouracil and Cisplatin) — At weeks 1, 5, 8 and 11
  * Day 1 to day 4: Fluorouracil 1 gr/m²/day
  * Day 1 or 2: Cisplatin 75 mg/m²

SUMMARY:
The scope of the trial is to predict the early complete clinical response to exclusive concomitant radiochemotherapy in esophageal cancer by the study of the pre- and per- therapeutic proteomic profile.

DETAILED DESCRIPTION:
Further informations will be provided by Centre Oscar Lambret.

ELIGIBILITY:
Inclusion Criteria:

* Invasive esophageal carcinoma at any stage (all T, N0 or N1, M0 or M1a), histologically proven
* Treated by exclusive concomitant radiochemotherapy
* Written informed consent

Exclusion Criteria:

* Presence of a second uncontrolled cancer
* Metastatic carcinoma
* Metastatic disease, except cervical lymphnodes... (M1a)
* In situ carcinoma
* Eso-gastric junction cancer (Siewert II ou III)
* Inclusion in a clinical trial with an experimental drug during the study and until 15 weeks after the end of radiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Proteomic analysis by Protein-Chip Technology of Ciphergen and mass spectrometry | 15 weeks after the end of irradiation
Initial complete clinical response | 15 weeks after the end of irradiation

SECONDARY OUTCOMES:
Prolonged clinical response at one year | One year after the end of irradiation

CONTACTS AND LOCATIONS:
Overall Officials: ADENIS Antoine, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (6):
- France (6):
  - Centre Paul Papin, Angers
  - Centre Hospitalier Universitaire, Brest
  - Centre François BACLESSE, Caen
  - Centre Oscar Lambret, Lille
  - Centre Eugène Marquis, Rennes
  - CHU - Hopital Charles Nicolle, Rouen